CLINICAL TRIAL: NCT01997515
Title: Ketamine Effect on Recovery and Respiratory Outcomes After Laparoscopic Gastric Reduction: A Randomized, Double-Blinded, Placebo Controlled Study
Brief Title: Ketamine Effect After Laparoscopic Gastric Reduction: A Randomized, Double-Blinded, Placebo Controlled Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Meltem Yilmaz, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00081191
Record Dates: First submitted 2013-11-18; First posted 2013-11-28 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Pain; Obesity; Hypoxia
Keywords: Quality of Recovery 40 Questionaire; Pain; Hypoxia; Gastric Surgery; Obesity; Ketamine
MeSH Terms: conditions — Pain; Obesity; Hypoxia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group K (Ketamine) (Active Comparator): Group K (ketamine) will receive 0.5mg /kg of ketamine bolus followed by an infusion of 0.5 mg/kg/hour of ketamine throughout the intraoperative period (Adjusted body weight).
  Interventions: Drug: Ketamine
- Group P (Placebo) (Placebo Comparator): Group P (placebo) will receive the same amount of saline.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ketamine — Group K (ketamine) will receive 0.5mg /kg of ketamine bolus followed by an infusion of 0.5 mg/kg/hour of ketamine throughout the intraoperative period (Adjusted body weight).
  Other Names: Ketalar
  Arms: Group K (Ketamine)
Drug: placebo — Group P (placebo) will receive the same amount of saline.
  Other Names: Sterile .9 Normal Saline
  Arms: Group P (Placebo)

SUMMARY:
Laparoscopic surgery for gastric reduction is frequently associated with high levels of postoperative pain. Postoperative pain is very often treated with opioids. However large doses of opioids can result in respiratory depression with hypoxemia especially in high risk patients with obstructive sleep apnea. since a large group of patients undergoing surgery for gastric reduction surgery also have obstructive sleep apnea, it is expected that these patients are also at high risk for postoperative respiratory depression and hypoxemia.

Intraoperative ketamine has been used as an effective multimodal agent to reduce postoperative pain. However, ketamine alone has not been examined to improve postoperative pain outcomes in patients undergoing gastric reduction surgery. More importantly, it is unknown if the use of intraoperative ketamine can lead to better overall quality of recovery in the same patient population. In addition, ketamine has been shown to improve ventilation but it remains to be determined if the intraoperative use of ketamine will result in less postoperative hypoxemic events.

The main objective of the current investigation is to examine the effect of intraoperative ketamine on postoperative quality of recovery after gastric reduction surgery. The investigators hypothesize that subjects receiving ketamine will have a greater global quality of recovery score than the ones receiving saline.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* surgery: laparoscopic gastric reduction (gastric sleeve or gastric bypass)
* ASA physical status classification I, II, III
* Body Mass Index >35kg/m2
* Fluent in English

Exclusion Criteria:

* History of allergy to protocol medications
* History of chronic opioid use
* Pregnant patients
* Drop out: Conversion to an open surgical route, patient or surgeon request.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Yilmaz, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han PY, Duffull SB, Kirkpatrick CM, Green B. Dosing in obesity: a simple solution to a big problem. Clin Pharmacol Ther. 2007 Nov;82(5):505-8. doi: 10.1038/sj.clpt.6100381. PMID 17952107

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group K (Ketamine) | Group P (Placebo)
Started | 40 | 40
Completed | 36 | 35
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group K (Ketamine) | Group P (Placebo) | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 27 | 62
  Male | 5 | 13 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery 40
Description: Scores on QOR (quality of recovery) 40 questionnaire. The QoR-40 score, which ranges from 40 to 200, representing very poor (low scores) to outstanding quality of recovery (high scores), respectively.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group K (Ketamine) | Group P (Placebo)
Number analyzed (Participants) | 36 | 35
score on a scale | 170 [158 to 177] | 179 [166 to 187]

2. Secondary Outcome: Postoperative Opioid Consumption
Description: Total number of opioids (morphine equivalents) consumed 24 hours after surgery
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: Morphine Equivalents
Arm/Group | Group K (Ketamine) | Group P (Placebo)
Number analyzed (Participants) | 36 | 35
Morphine Equivalents | 4.45 [3 to 7.83] | 6.3 [3.6 to 10.1]

3. Secondary Outcome: Postoperative Pain Scores
Description: Participants pain scores will be recorded at 24 hours after surgery. Pain scores range from 0 (no pain) to 10 (worst pain imaginable).
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group K (Ketamine) | Group P (Placebo)
Number analyzed (Participants) | 36 | 35
score on a scale | 4 [2.25 to 5.75] | 4 [2 to 5]

4. Secondary Outcome: Length of Hospital Stay
Description: The subjects length of hospital stay will be recorded. Length of stay is defined as day of surgery to date of discharge from the hospital which may be up to 2 weeks..
Time Frame: Up to 2 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group K (Ketamine) | Group P (Placebo)
Number analyzed (Participants) | 36 | 35
days | 2.00 [2.00 to 2.75] | 2.00 [2.00 to 2.00]

ADVERSE EVENTS:
Time Frame: Time period for adverse events were collected was until discharge from hospital which is indefinite but generally up to 2 weeks.
Arm/Group | Group K (Ketamine) | Group P (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT01997515/Prot_SAP_000.pdf